CLINICAL TRIAL: NCT03029832
Title: A Phase II, Multicenter, Randomized, Placebo-Controlled, Double-Blind Study of MOXR0916 in Combination With Atezolizumab Versus Atezolizumab Alone in Patients With Untreated Locally Advanced or Metastatic Urothelial Carcinoma Who Are Ineligible for Cisplatin-Based Therapy
Brief Title: A Study of MOXR0916 in Combination With Atezolizumab Versus Atezolizumab Alone in Participants With Untreated Locally Advanced or Metastatic Urothelial Carcinoma Who Are Ineligible for Cisplatin-Based Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was prematurely terminated due to slow patient accrual and discontinuation of clinical development of MOXR0916 due to Sponsor's strategic priorities.
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO39590; 2016-004165-58 (EudraCT Number)
Record Dates: First submitted 2017-01-18; First posted 2017-01-24 (Estimated); Results first posted 2019-05-31 (Actual); Last update posted 2019-05-31 (Actual); Status verified 2019-05

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — atezolizumab

STUDY DESIGN:
Masking Description: The study design has been amended in that the study blinding will not be maintained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MOXR0916 plus Atezolizumab (Experimental)
  Interventions: Drug: MOXR0916; Drug: Atezolizumab
- Atezolizumab (Active Comparator)
  Interventions: Drug: Atezolizumab

INTERVENTIONS:
Drug: MOXR0916 — MOXR0916, 300 milligram (mg) by intravenous (IV) infusion on Day 1 of each 21-day cycle.
  Arms: MOXR0916 plus Atezolizumab
Drug: Atezolizumab — Atezolizumab, 1200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle.

SUMMARY:
This is a Phase II, multicenter, randomized, placebo-controlled, double-blind study to evaluate the safety and efficacy of MOXR0916 in combination with atezolizumab versus placebo and atezolizumab in participants with locally advanced or metastatic urothelial carcinoma (UC) who have not received prior systemic therapy in the locally advanced/metastatic setting and who are ineligible to receive cisplatin-based therapy.

DETAILED DESCRIPTION:
The study design has been amended after the decision to prematurely stop patient accrual due to enrollment challenges. As only 5 participants were enrolled, the study blinding will not be maintained, and placebo infusions will not be administered. Patients assigned to the MOXR0916 arm may continue study treatment with the combination of atezolizumab and MOXR0916 or with atezolizumab alone based on a discussion of benefit and risk with the treating investigator.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of <= 2
* Life expectancy >= 12 weeks
* Histologically or cytologically confirmed locally advanced or metastatic urothelial carcinoma (UC)
* Availability of a representative formalin-fixed paraffin-embedded tumor specimen
* No prior systemic therapy for inoperable locally advanced or metastatic UC
* Ineligible for cisplatin-based chemotherapy as defined by any one of the following criteria: Impaired renal function (glomerular filtration rate [GFR] > 30 but < 60 milliliter/minute [mL/min]); National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version (v) 4.0 Grade >= 2 audiometric hearing loss (of 25 Decibel at two contiguous frequencies or more severe); NCI CTCAE v 4.0 Grade >= 2 peripheral neuropathy; ECOG Performance Status of 2
* Measurable disease according to Response Evaluation Criteria in Solid Tumors v1.1
* Adequate hematologic and end-organ function

Exclusion Criteria:

* Significant cardiovascular disease
* Known clinically significant liver disease
* Any approved anti-cancer therapy, including chemotherapy or hormonal therapy, within 3 weeks prior to initiation of study treatment
* Prior treatment with CD137 or OX40 agonists, anti-cytotoxic T-lymphocyte-associated protein (CTLA4), anti-programmed death-1 (PD-1), anti- programmed death-ligand 1 (PD-L1), anti-CD-27, anti- glucocorticoid-induced tumor necrosis factor receptor (GITR) therapeutic antibody or pathway-targeting agents
* Untreated central nervous system (CNS) metastases or active (progressing or requiring corticosteroids for symptomatic control) CNS metastases
* Any history of leptomeningeal disease
* Malignancies other than UC within 5 years prior to Cycle 1, Day 1
* History of autoimmune disease
* History of idiopathic pulmonary fibrosis, pneumonitis, organizing pneumonia, or evidence of active pneumonitis on screening chest computed tomography scan
* Active hepatitis B and C virus infection
* Positive HIV test at screening
* Active tuberculosis
* Prior allogeneic stem cell or solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-04-27 (Actual); Primary Completion 2018-04-25 (Actual); Study Completion 2018-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (22):
- United States (15):
  - Arizona Oncology - HOPE Wilmot, Tucson, Arizona
  - University of Colorado, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - Miami Cancer Institute of Baptist Health, Inc., Miami, Florida
  - University of Chicago; Hematology/Oncology, Chicago, Illinois
  - Kansas City - Menorah Medical Center, Kansas City, Kansas
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Nebraska Methodist Hospital; Cancer Center, Omaha, Nebraska
  - New York Oncology Hematology, P.C., Albany, New York
  - Columbia University Medical Center; Clinical Research Management Office, New York, New York
  - Onc/Hem Care Clin Trials LLC, Cincinnati, Ohio
  - SCRI Tennessee Oncology Chattanooga, Chattanooga, Tennessee
  - Sarah Cannon Research Inst., Nashville, Tennessee
  - Texas Oncology-Baylor Sammons Cancer Center, Dallas, Texas
  - Virginia Oncology Associates - Lake Wright Cancer Center, Norfolk, Virginia
- GasthuisZusters Antwerpen, Wilrijk, Belgium
- Princess Margaret Cancer Center, Toronto, Ontario, Canada
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center - Oncology, Seoul
- United Kingdom (2):
  - Leicester Royal Infirmary NHS Trust, Leicester
  - Barts and the London NHS Trust., London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MOXR0916 Plus Atezolizumab: Participants were administered MOXR0916, 300 milligram (mg) and atezolizumab, 1200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle.
- Atezolizumab: Participants were administered atezolizumab, 1200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle.
Period: Overall Study
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Started | 4 | 1
Completed | 0 | 0
Not Completed | 4 | 1
Not completed — Safety Follow-Up Completed | 2 | 0
Not completed — Death due to Disease Progression | 1 | 0
Not completed — Study Terminated By Sponsor | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab | Total
Number analyzed (Participants) | 4 | 1 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 3 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 1 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first. Per RECIST v1.1, progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum of diameters on study (including baseline); and an absolute increase of >= 5 millimeter (mm) in the sum of diameters.
Time Frame: Up to approximately 45 months
Population: Due to early termination, no formal analyses were performed for PFS.
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Overall Survival (OS)
Description: Kaplan Meier estimate of median OS was defined as the time at which half of the participants had died, regardless of the cause of death.
Time Frame: Up to approximately 45 months
Population: Due to early termination, no formal analyses were performed for OS.
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Objective Response (OR) According to RECIST v1.1
Description: OR is defined as a complete response (CR) or partial response (PR) on two consecutive occasions >= 4 weeks apart, as determined by the investigator according to RECIST v1.1. CR is defined as the disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: Up to approximately 45 months
Population: Due to early termination, no formal analyses were performed for OR.
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Duration of Objective Response (DOR) According to RECIST v1.1
Description: DOR is defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause, whichever occurs first, as determined by the investigator according to RECIST v1.1. Objective response is defined as a complete response (CR) or partial response (PR) on two consecutive occasions ≥ 4 weeks apart. CR is defined as the disappearance of all target lesions. PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: Up to approximately 45 months
Population: Due to early termination, no formal analyses were performed for DOR.
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Pain Progression, Pain Palliation, and Fatigue Progression as Measured by Participant-Reported Severity According to the M. D. Anderson Symptom Inventory (MDASI)
Description: The MDASI is a cancer-related, self-reported questionnaire consisting of 19 items assessing symptom severity and interference with different aspects of a participant's life. The MDASI items are rated from 0 to 10, with 0 indicating that the symptom is either not present or does not interfere with the participant's activities and 10 indicating that the symptom is "as bad as you can imagine" or "interfered completely" with the participant's life.
Time Frame: Up to approximately 45 months
Population: Due to early termination, no formal analyses were performed for time to pain progression, pain palliation and fatigue progression.
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Percentage of Participants Reporting Symptom Interference With Daily Living at the Time of Progression According to the MDASI
Description: as for outcome 5
Time Frame: Up to approximately 45 months
Population: Due to early termination, no formal analyses were performed for percentage of participants reporting symptom interference with daily living at the time of progression according to the MDASI
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants With Adverse Event (AEs)
Description: An adverse event is any untoward medical occurrence, regardless of causal attribution.
Time Frame: Up to approximately 45 months
Population: The safety population was defined as all participants who have received at least one dose of study medication. Data were collected but are not being summarized due to privacy concerns with the low number of patients analyzed.
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Area Under the Plasma Drug Concentration-time Curve (AUC) of MOXR0916 and Atezolizumab
Description: AUC represents the body's exposure to an administered drug.
Time Frame: Cycle 1 (each cycle is 21 days), Day 1: predose and 30 min. after atezolizumab infusion; Cycle 1, on Days 8 and 15. Cycles 2 4, Day 1: predose and 30 min. after atezolizumab infusion. Cycles 8, 12, and 16: predose
Population: Due to early termination, no formal analyses were performed for any of the pharmacokinetic measures.
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Maximum Plasma Concentration (Cmax) of MOXR0916 and Atezolizumab
Description: Cmax refers to the maximum (or peak) serum concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and prior to the administration of a second dose.
Time Frame: as for outcome 8
Population: Due to early termination, no formal analyses were performed for any of the pharmacokinetic measures.
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Minimum Plasma Concentration (Cmin) of MOXR0916 and Atezolizumab
Description: Cmin refers to the minimum (trough) serum concentration of a drug in a specified compartment or test area of the body.
Time Frame: as for outcome 8
Population: Due to early termination, no formal analyses were performed for any of the pharmacokinetic measures.
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Clearance of MOXR0916 and Atezolizumab
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes.
Time Frame: as for outcome 8
Population: Due to early termination, no formal analyses were performed for any of the pharmacokinetic measures.
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to MOXR0916 and Atezolizumab
Description: ATAs may be produced by the body in response to an administered drug.
Time Frame: Cycles 1 - 4 and 8, 12, and 16 (each cycle is 21 days), Day 1: predose
Population: Due to early termination, no formal analyses were performed for percentage of participants with ATAs to MOXR0916 and Atezolizumab.
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 45 months
Description: The safety population is defined as all patients who received at least one dose of the study medication. Data were collected for the adverse events but are not being summarized due to privacy concerns with low number of patients analyzed.
Arm/Group | MOXR0916 Plus Atezolizumab | Atezolizumab
All-Cause Mortality (participants affected / at risk) | 1/4 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT03029832/Prot_SAP_000.pdf